CLINICAL TRIAL: NCT04992702
Title: The Effect of a Brief, Web-Based Animated Video for Improving Comprehension and Implementation Feasibility for Reducing Anterior Cruciate Ligament Injury: A Three-Arm Randomized Controlled Trial
Brief Title: Effect of Animated Video on Comprehension and Implementation Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan Technological University (Other)
Responsible Party: Principal Investigator, Erich Petushek, Assistant Professor, Michigan Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1521444-1
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: multimedia; education; information; knee; coach; learning
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animated Video (Experimental): The information in the ACL animated video (https://vimeo.com/281721823) was displayed as a story of a typical athlete who sustained an injury and how this could be prevented through evidence-based prevention strategies.
  Interventions: Behavioral: Animated Video
- Web-based Article (Active Comparator): The active control group received commonly accessed information from a WebMD web-based article on ACL injury prevention.
  Interventions: Behavioral: Animated Video
- Placebo control (Placebo Comparator): The placebo control group intervention received an educational video from the CDC about concussions that is comparable in duration to that of the ACL video (https://youtu.be/fSRWF44wgn8).
  Interventions: Behavioral: Animated Video

INTERVENTIONS:
Behavioral: Animated Video — Animated video to improve learning and motivation
  Other Names: Multimedia video

SUMMARY:
The aim of this study is to evaluate the effects of a brief web-based educational intervention on improving Anterior Cruciate Ligament (ACL) injury prevention comprehension and implementation feasibility among coaches of athletes participating in landing and cutting sports (e.g., soccer, basketball, football, etc.). The two main hypotheses are that, compared to both an active and placebo control group, the brief animated video will produce greater improvements in:

1. Overall comprehension of ACL injury risk and mitigation: placebo control group < active control group < intervention group.
2. Feasibility of utilizing ACL injury prevention strategies: placebo control group < active control group < intervention group.

Exploratory hypothesis: The brief animated video will produce greater improvements in various subcomponents of comprehension-specifically: basic ACL knowledge, risk knowledge, prevention knowledge and severity knowledge compared to both active and placebo control group conditions.

DETAILED DESCRIPTION:
This study is a computer-based, three-arm pre-post randomized control design trial. Participants were randomized into an intervention group, active control group or passive control group on a 1:1:1 ratio by a computer-generated algorithm embedded within the Qualtrics software (Qualtrics, Provo, UT). Sports coaches of youth and adolescent athletes in various landing and cutting sports (e.g., soccer, basketball, volleyball, etc.) in the United States were recruited and invited through Qualtrics' panelists. The intervention group was shown a three-minute animated video consisting of various information components aimed at improving capability, motivation and opportunity to implement ACL injury prevention strategies. The active control group received commonly accessed information from a WebMD web-based article on ACL injury prevention. The placebo control group intervention received an educational video from the CDC about concussions that is comparable in duration to that of the ACL video. Overall ACL comprehension-composed of basic ACL knowledge, risk knowledge, prevention knowledge, and severity knowledge-as well as implementation feasibility were all measured prior to and immediately following the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Sports coaches of youth and adolescent athletes in various landing and cutting sports (e.g., soccer, basketball, volleyball, etc.) in the United States.

Exclusion Criteria:

* Non sport coach or coach of non-landing and cutting sport (e.g., golf, swimming).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Overall anterior cruciate ligament injury comprehension percent correct | Immediately following intervention
  Items that measure ACL knowledge were gathered from peer reviewed, published articles. The scale consisted of 15 multiple choice items that assessed individuals knowledge about diverse issues with ACL injury such as risk, prevention, and consequences of the injury.

SECONDARY OUTCOMES:
Average implementation feasibility measured by the feasibility of the intervention scale | Immediately following intervention
  The feasibility of the intervention measure was used to assess the likelihood that the coach would successfully implement evidence-based prevention strategies. The 4 items consisted of the root phrase: "An ACL injury prevention program seems" followed by (1) implementable, (2) possible, (3) doable and (4) easy to use. The items were rated on a 5-point Likert scale ranging from completely disagree to completely agree. The average of the 4 items was used for the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Technological University, Houghton, Michigan, United States

IPD SHARING:
Plan to Share IPD: No